CLINICAL TRIAL: NCT01652742
Title: Pharmacokinetics and Pharmacodynamics of BI 135585 XX Administered as Oral Dose in Healthy Male Volunteers (Open-label, Single-dose Trial)
Brief Title: Study to Explore Pharmacokinetics and Pharmacodynamics of a Single Rising Dose of BI 135585 XX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1283.34; 2012-000844-85 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Healthy

ARMS (1):
- BI 135585 XX (Experimental): one single dose
  Interventions: Drug: BI 135585 XX

INTERVENTIONS:
Drug: BI 135585 XX — one single dose

SUMMARY:
To investigate the pharmacokinetics and pharmacodynamics of BI 135585 XX following single dose administration.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects
2. overweight or obese

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 4 days postdose
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 4 days postdose

SECONDARY OUTCOMES:
AUC0-8 of BI 135585 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 4 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1283.34.1 Boehringer Ingelheim Investigational Site, Neuss, Germany